CLINICAL TRIAL: NCT01089088
Title: A Phase II Single-Arm Trial to Evaluate Cisplatin and Gemcitabine Chemotherapy in Combination With Sunitinib for First-Line Treatment of Patients With Advanced Transitional Carcinoma of the Urothelium
Brief Title: Gemcitabine Hydrochloride, Cisplatin, and Sunitinib Malate as First-Line Therapy in Treating Patients With Locally Advanced And/or Metastatic Transitional Cell Carcinoma of the Urothelium (SUCCINCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Principal Investigator, Lisette Nixon, Senior Trial Manager, Cardiff University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000667764; WCTU-SUCCINCT; ISRCTN54607216; EUDRACT-2007-007591-42; EU-21013; WCTU-SPON-416-07; CRUK-07/044
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2013-02

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent urethral cancer; recurrent transitional cell cancer of the renal pelvis and ureter; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; transitional cell carcinoma of the bladder; stage IV bladder cancer; recurrent bladder cancer; anterior urethral cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Cisplatin; Sunitinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin — Up to six 21 day chemotherapy cycles:
  Cisplatin 70mg/m2 (IV day 1) Gemcitabine 1000mg/m2 (IV days 1 & 8) Sunitinib 37.5mg (po days 2 to 15)
  Other Names: Sutent
Drug: gemcitabine hydrochloride — Up to six 21 day chemotherapy cycles:
  Cisplatin 70mg/m2 (IV day 1) Gemcitabine 1000mg/m2 (IV days 1 & 8) Sunitinib 37.5mg (po days 2 to 15)
Drug: sunitinib malate — Up to six 21 day chemotherapy cycles:
  Cisplatin 70mg/m2 (IV day 1) Gemcitabine 1000mg/m2 (IV days 1 & 8) Sunitinib 37.5mg (po days 2 to 15)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving gemcitabine hydrochloride and cisplatin together with sunitinib malate may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving gemcitabine hydrochloride and cisplatin together with sunitinib malate and to see how well it works as first-line therapy in treating patients with locally advanced and/or metastatic transitional cell carcinoma of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the activity, safety, and feasibility of gemcitabine hydrochloride and cisplatin in combination with sunitinib malate as first-line therapy in patients with locally advanced and/or metastatic transitional carcinoma of the urothelium.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, cisplatin IV over 3-4 hours on day 1, and oral sunitinib malate once daily on days 2-15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 6 months and 1 year.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the urothelium

  * Pure or mixed histology
  * Upper or lower urinary tract
* Radiologically measurable, locally advanced and/or metastatic disease not amenable to curative treatment with surgery or radiotherapy meeting 1 of the following criteria:

  * T4b (bladder) or T4 (renal pelvis/ureter), any N, any M
  * Any T, N2-3, any M
  * Any T, any N, M1
* No urothelial cancer for which subsequent radical treatment is being considered with a view to possibly cure the disease
* No history of CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and ALP ≤ 2.5 times ULN
* GFR ≥ 60 mL/min (uncorrected for surface area and measured by isotopic means)
* PT or INR ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Fit to receive cisplatin-containing combination chemotherapy
* No previous malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix, or incidental localized prostate cancer
* No known HIV positivity or chronic hepatitis B or C infection
* No uncontrolled hypertension
* No symptomatic coronary artery disease, myocardial infarction within the past 6 months, congestive cardiac failure (NYHA class III-IV disease), or uncontrolled or symptomatic cardiac arrhythmia
* No clinically significant bacterial or fungal infection
* No concurrent grapefruit juice

PRIOR CONCURRENT THERAPY:

* At least 1 month since prior radiotherapy or radiotherapy involving more than 30% of total bone marrow volume
* At least 1 month since prior investigational drug
* No prior systemic therapy for locally advanced or metastatic disease

  * Patients who have received prior neoadjuvant or adjuvant chemotherapy for urothelial cancer (up to 4 courses), completed at least 6 months prior to first documented disease progression, are eligible
* No concurrent anticoagulant therapy with warfarin or unfractionated heparin

  * Patients requiring anticoagulation may be entered on study after successful conversion to low molecular weight heparin
* No concurrent medications that have known adverse interactions with sunitinib malate (i.e., strong CYP3A4 inhibitors or inducers)
* No prior or concurrent live vaccines (e.g., measles, mumps, rubella, oral polio, bacille Calmette-Guérin [BCG], yellow fever, varicella, and TY21a typhoid vaccines)

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  Proportion of patients progression free at 6 months

SECONDARY OUTCOMES:
Toxicity during and after treatment according to NCI CTCAE v 3.0 | 1 Year
Tolerability (side effects) and feasibility of use (number of patients requiring dose delays or reduction and/or treatment withdrawal) | 1 year
Overall survival | 3 years
Progression-free survival (time-to-event) | 1 year
Objective (radiological) response rate according to RECIST | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tom Geldart, Principal Investigator — Royal Bournemouth Hospital
Locations (16):
- United Kingdom (16):
  - Bristol Haematology and Oncology Centre, Bristol, Avon
  - Castle Hill Hospital, Cottingham, East Yorkshire
  - Royal Bournemouth Hospital, Bournemouth, England
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - The Royal Marsden Hospitals (Surrey), Sutton, Surrey
  - St James's University Hospital, Leeds, Yorkshire
  - Addenbrooke's Hospital, Cambridge
  - Velindre Hospital, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St Bartholomew's Hospital, London
  - Hammersmith Hospital, London
  - St Mary's Hospital (Paddington), London
  - Charing Cross Hospital, London
  - Christie Hospital, Manchester
  - Southampton General Hospital, Southampton

REFERENCES:
- [Result] Chang SS. Re: SUCCINCT: An Open-Label, Single-Arm, Non-Randomised, Phase 2 Trial of Gemcitabine and Cisplatin Chemotherapy in Combination with Sunitinib as First-Line Treatment for Patients with Advanced Urothelial Carcinoma. J Urol. 2015 Dec;194(6):1583-4. doi: 10.1016/j.juro.2015.09.005. Epub 2015 Sep 5. No abstract available. PMID 26582660
- See also: Summary on sponsor website — https://www.cardiff.ac.uk/centre-for-trials-research/research/studies-and-trials/view/succinct
- See also: Trial Publication link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4410296/